CLINICAL TRIAL: NCT05591235
Title: Effect of Metformin, Dapagliflozin, Fixed Combination of Metformin and Pioglitazone in Overweighted Patients With Newly Diagnosed Type 2 Diabetes
Brief Title: Effect of Metformin, Dapagliflozin, Combination of Metformin and Pioglitazone in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20220314-01
Record Dates: First submitted 2022-10-16; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-09

CONDITIONS: Type2diabetes; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Metformin; dapagliflozin; Pioglitazone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metformin (Active Comparator)
  Interventions: Drug: Dapagliflozin; Drug: Fixed-dose combination of metformin and pioglitazone (500mg metformin plus 15mg pioglitazone)
- Fixed-dose combination of metformin and pioglitazone (500mg metformin plus 15mg pioglitazone) (Active Comparator)
  Interventions: Drug: Metformin; Drug: Dapagliflozin
- Dapagliflozin (Active Comparator)
  Interventions: Drug: Metformin; Drug: Fixed-dose combination of metformin and pioglitazone (500mg metformin plus 15mg pioglitazone)

INTERVENTIONS:
Drug: Metformin — After the screening period, eligible subjects took the hyperinsulinemic euglycemic clamp test and were then admitted to insulin with metformin for 4 weeks. During this timeframe, all patients were instructed to change the insulin pump infusion site and provide one profile of 7-point self-monitored blood glucose every three days. The insulin doses were titrated every day by physicians to achieve the glycemic goal. Participants who failed to attain the glycemic target in three consecutive times or could not afford the side effects of hypoglycemic medications were excluded from this study. On the last day of week 4, a FreeStyle Libre Pro Sensor (FGM system) was inserted to record the glycemic data for up to 14 days. At the end of week 5, all antidiabetic agents were stopped and the hyperinsulinemic euglycemic clamp test was performed again for remaining subjects.
  Arms: Dapagliflozin; Fixed-dose combination of metformin and pioglitazone (500mg metformin plus 15mg pioglitazone)
Drug: Dapagliflozin — After the screening period, eligible subjects took the hyperinsulinemic euglycemic clamp test and were then admitted to insulin with dapagliflozin (100mg one day) for 4 weeks. During this timeframe, all patients were instructed to change the insulin pump infusion site and provide one profile of 7-point self-monitored blood glucose every three days. The insulin doses were titrated every day by physicians to achieve the glycemic goal. Participants who failed to attain the glycemic target in three consecutive times or could not afford the side effects of hypoglycemic medications were excluded from this study. On the last day of week 4, a FreeStyle Libre Pro Sensor (FGM system) was inserted to record the glycemic data for up to 14 days. At the end of week 5, all antidiabetic agents were stopped and the hyperinsulinemic euglycemic clamp test was performed again for remaining subjects.
  Arms: Fixed-dose combination of metformin and pioglitazone (500mg metformin plus 15mg pioglitazone); Metformin
Drug: Fixed-dose combination of metformin and pioglitazone (500mg metformin plus 15mg pioglitazone) — After the screening period, eligible subjects took the hyperinsulinemic euglycemic clamp test and were then admitted to insulin with fixed-dose combination of metformin and pioglitazone (two tablets of 500mg metformin plus 15mg pioglitazone) for 4 weeks. During this timeframe, all patients were instructed to change the insulin pump infusion site and provide one profile of 7-point self-monitored blood glucose every three days. The insulin doses were titrated every day by physicians to achieve the glycemic goal. Participants who failed to attain the glycemic target in three consecutive times or could not afford the side effects of hypoglycemic medications were excluded from this study. On the last day of week 4, a FreeStyle Libre Pro Sensor (FGM system) was inserted to record the glycemic data for up to 14 days. At the end of week 5, all antidiabetic agents were stopped and the hyperinsulinemic euglycemic clamp test was performed again for remaining subjects.
  Arms: Dapagliflozin; Metformin

SUMMARY:
Although, a number of drugs are promising treatment strategies for insulin resistance, a critical question arises to which drug benefits patients with type 2 diabetes more from reduced insulin resistance and consequent glycemic control. In this study, we aim to evaluate the effect of metformin, dapagliflozin and the fixed-dose combination of metformin and pioglitazone (500mg metformin plus 15mg pioglitazone) on insulin sensitivity and glycemic control in overweight patients with newly diagnosed type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in this present study;
* Regular diet and exercise;
* Age 18 to 60 years;
* Screening glycated hemoglobin (HbA1c) > 9.0%;
* Body mass index (BMI) ≥ 24.0 kg/m2

Exclusion Criteria:

* Other forms of diabetes;
* Insulin allergy or intolerance of metformin, pioglitazone and dapagliflozin;
* Renal dysfunction (estimated glomerular filtration rate < 45 mL/min);
* Severe liver disease or elevated transaminases (2.5-fold the upper limit);
* History of alcohol dependence or drug abuse in the past 5 years;
* Systemic steroids therapy or other medication influencing cholesterol metabolism in the past 3 months;
* Acute infection or stress state 1 month prior to this study;
* Pregnancy or lactation;
* History of diabetic ketoacidosis (DKA) within the previous year;
* Psychiatric disease;
* Other comorbid serious condition including severe heart and pulmonary disease, heart failure of New York Heart Association class IV, and tumors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | week 5
  change from baseline insulin resistance at the fifth week

IPD SHARING:
Plan to Share IPD: No